CLINICAL TRIAL: NCT04760808
Title: Evaluation of Cerebrospinal Fluid Flow by MRI in Adolescent Idiopathic Scoliosis, From Its Signaling Through the Study of Trunk Graviception and Proprioception
Brief Title: Evaluation of Cerebrospinal Fluid Flow in Adolescent Idiopathic Scoliosis
Acronym: MEDULLOSCOL
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: SSR pédiatrique Marc Sautelet (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC-P0093
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: cerebrospinal fluid flow; MRI; Graviception; Postural control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIS group
  Interventions: Diagnostic Test: Baseline Clinical Examination; Radiation: Initial 3T MRI of the Brain and Spine; Diagnostic Test: 6-month Follow-up Clinical Examination; Radiation: 6-month Follow-up 3T MRI of the Brain and Spine
- Control Group
  Interventions: Diagnostic Test: Baseline Clinical Examination; Radiation: Initial 3T MRI of the Brain and Spine

INTERVENTIONS:
Diagnostic Test: Baseline Clinical Examination — Evaluations of Postural control; Subjective postural vertical; Subjective visual vertical; Verticality perception
Radiation: Initial 3T MRI of the Brain and Spine — Non-injected CSF flow MRI
Diagnostic Test: 6-month Follow-up Clinical Examination — Evaluations of Postural control; Subjective postural vertical; Subjective visual vertical; Verticality perception
  Groups: AIS group
Radiation: 6-month Follow-up 3T MRI of the Brain and Spine — Non-injected CSF flow MRI
  Groups: AIS group

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is the most frequent spinal deformity in adolescence, but its etiology remains unknown. Recent publications suggest a link between ciliopathy and AIS. More specifically a modification of the cerebro-spinal fluid (CSF) flow by ciliary dysfunction could be at the origin of a scoliotic deformity.

This study aims to compare the CSF flow measured by magnetic resonance imaging (MRI) in an AIS group and a control group.

ELIGIBILITY:
Common Inclusion Criteria for the 2 groups :

* Female subject aged 12 to < 18 years old
* Affiliated to the French social security system
* Having signed the inform consent form
* Whose parents have given their consent

Additional Inclusion Criteria for the AIS group:

* Subject with right thoracic AIS defined by the existence of a 3D spine deformation with a frontal deviation to right dorsal convexity with a Cobb angle of at least 20°, and a rotation of at least 20°, as evidenced by the presence of a vertebral gibbosity ≥ 5° at the Bunnel scoliometer.

If the scoliosis has more than one curvature, the right chest curvature should be the greatest high (highest frontal Cobb angle)

* Subject with x-rays of total spine, face and profile under load, according to the EOS technique, dating from less than 3 months.

Common Exclusion Criteria for the 2 groups:

* Instability to submit to the medical follow-up of the study for psychic, social or geographical reasons
* At least 6 "cafe au lait" spots with a size ≥ 1.5 cm (may be suggestive of neurofibromatosis)
* Ligament hyperlaxity confirmed by a Beighton score >4/9 (which may be suggestive of scoliosis secondary)
* Contraindications of a cerebro-medullary MRI: claustrophobia, foreign bodies, and ferrometallic clips of the trunk or cephalic segment, cochlear implants, stimulators and implantable cardiac defibrillators, insulin pump
* Inequality in length of the lower limbs ≥ 20 mm on clinical examination
* Subject presenting neurological signs (signs of pyramidal irritation, sensory-motor deficit, clinical signs suggestive of cerebellar pathology ...)
* Known vestibular pathology
* Taking psychotropic drugs

Additional exclusion criterion for the AIS group:

* Subject with secondary scoliosis : neurological, orthopedic, malformative...

Additional criteria for the control group:

* Subject with a scoliosis angle ≥ 10° on a photogrammetric screening assessment (optical process, non-irradiating, which allows an Morphometric evaluation of the trunk in 3D, thanks to the analysis of the trunk reliefs)
* Subject whose clinical examination shows a gibbosity measurable (>5°) with the scoliometer of Bunnel

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 2 Groups:
  * 35 cases: Female Adolescents with AIS
  * 35 controls: Female subjects without scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
CSF flow (cm/s) at the 7th thoracic vertebra (T7) | 6 months
  The flow will be measured by MRI

SECONDARY OUTCOMES:
CSF flow (cm/s) at the cervico-occipital junction | 6 months
  The flow will be measured by MRI
CSF flow (cm/s) at the cerebral aqueduct | 6 months
  The flow will be measured by MRI
Prevalence of spinal cord abnormalities | 6 months
  Measured by MRI
Correlation between the Body Mass Index and the CSF flow (cm/s) at the 7th thoracic vertebra (T7) | 6 months
  This association will be studied by a linear regression analysis
Cobb frontal angle in degrees | 6 month
  The measurement of radiographic parameters will be done with the EOS system. The EOS system is a new slot-scanning radiological device that allows simultaneous acquisition of frontal and lateral images. It is composed of two X-ray sources, shaped as fan beams through collimation slits.
Distance between the vertical line passing through the middle of the sacrum and the vertical line passing through the spine of the 7th cervical vertebra. | 6 month
Angle of thoracic kyphosis T4-T12 in degrees | 6 months
  The measurement of radiographic parameters will be done with the EOS system.
Lumbar lordosis angle L1-L5 in degrees | 6 months
  The measurement of radiographic parameters will be done with the EOS system.
Lumbo-sacral angle L5-S1 in degrees | 6 months
  The measurement of radiographic parameters will be done with the EOS system The measurement of radiographic parameters will be done with the EOS system.
Pelvic incidence in degrees | 6 months
  The measurement of radiographic parameters will be done with the EOS system
Subjective Postural Vertical Measurement in degrees | 6 months
Subjective Visual Vertical Sight Measurement in degrees | 6 months
Proprioception Measurement in degrees | 6 months
  Proprioception measurement obtained by trunk repositioning error test (Formetric system)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François CATANZARITI, MD, Principal Investigator — SSR Marc Sautelet, France
Locations (2):
- France (2):
  - SSR Pédiatrique Marc Sautelet, Villeneuve-d'Ascq, Nord (59)
  - GHICL Hôpital Saint Philibert, service d'Imagerie Médicale, Lomme, Nord

IPD SHARING:
Plan to Share IPD: No